CLINICAL TRIAL: NCT03612882
Title: Investigating the Relationship Between Sedentary Behaviour and Subjective Well-being in University Students: A Cross-sectional Study
Brief Title: Sedentary Behaviour and Subjective Well-being
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 111662
Record Dates: First submitted 2018-07-23; First posted 2018-08-02 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2019-09

CONDITIONS: Sedentary Behaviour
Keywords: Sedentary Behaviour; Subjective Well-Being; University Students

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Western University Students: Online questionnaire
  Interventions: Other: Online questionnaire

INTERVENTIONS:
Other: Online questionnaire — Online questionnaire assessing sedentary behaviour, physical activity, subjective well-being, life satisfaction, depression, anxiety, and demographics

SUMMARY:
This study will investigate the relationship between sedentary behaviour and subjective well-being among a sample of university students. Eligible participants will fill out an online survey with questions assessing their sedentary behaviour, physical activity, subjective well-being, life satisfaction, depression, anxiety, and demographic variables.

DETAILED DESCRIPTION:
An electronic survey will be used to assess outcomes of interest (i.e., demographics, sedentary behaviour and physical activity history, subjective well-being, life satisfaction, depression, and anxiety). The survey will be created and hosted on SoSci Survey. Interested participants will contact the investigators and will be sent a personal link to access the survey. Upon following the link, participants will answer inclusion/exclusion criteria and give electronic consent. Upon confirming consent and eligibility, participants will complete the survey. Upon completion of the survey, participants will be thanked and offered an entry into a draw.

ELIGIBILITY:
Inclusion Criteria:

* Currently a full-time student enrolled at Western University
* Are 18 years of age or older
* Are able to read and write in English
* Have access to a computer with internet

Exclusion Criteria:

* Part-time enrollment or currently on a leave of absence from full-time studies at Western University

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Full-time University students attending Western University
Sampling Method: Non-Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Subjective Well-Being (Affect) | Baseline
  Subjective Well-Being (specifically, affect) will be assessed through the Positive Affect & Negative Affect Scale (PANAS).
  The PANAS consists of a number of words that describe different feelings and emotions. Participants indicate the extent to which they feel a particular feeling and emotion over the past week, using a 5-point scale that ranges from 1 "very slightly or not at all" to 5 "extremely".
  An overall score for both positive and negative affect is calculated by summing up the points for those particular feelings/emotions (e.g., interested for positive affect, distressed for negative affect). Scores for positive affect can range from 10-50, with higher scores representing higher levels of positive affect. Scores for negative affect can range from 10-50, with lower scores representing lower levels of negative affect.
Subjective Well-Being (Life Satisfaction) | Baseline
  Subjective Well-Being (specifically, life satisfaction) will be assessed through the Satisfaction with Life Scale (SWLS); a 5-item scale designed to measure global cognitive judgments of one's life satisfaction.
  Participants indicate how much they agree or disagree with each of the 5-items over the past week, using a 7-point scale that ranges from 7 "strongly agree" to 1 "strongly disagree". An overall score (from 5 to 35) is calculated through summing the responses to the 5-items.
  Recommended cutoffs for interpretation are: 5-9, extremely dissatisfied; 10-14, dissatisfied; 15-19, slightly dissatisfied; 20, neutral; 21-25, slightly satisfied; 26-30, satisfied; 31-35, very satisfied.
Subjective Well-Being | Past seven days
  Subjective Well-Being will be assessed through the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS).
  The WEMWBS consists of 14-items that assesses subjective well-being through both hedonic and eudaimonic dimensions of well-being. Participants select the option that best describes their experience with each of the 14-items over the last week (note: the original questionnaire assesses the last two weeks), using a 5-point scale that ranges from 1 "none of the time" to 5 "all of the time".
  A total score is calculated by summing the 14 individual statement scores. The minimum score is 14 and the maximum is 70, with higher scores indicating greater levels of subjective well-being.

SECONDARY OUTCOMES:
Physical Activity | Past seven days
  Average total weekday and weekend time spent in moderate and vigorous physical activities in the last 7 days will be assessed through the International Physical Activity Questionnaire Seven - Short Form Past 7 Days (IPAQ-S7S).
  Participants report how many days per week (0-7) and how many hours/minutes per day they spent engaged in vigorous and moderate intensity physical activity, as well as walking.
Sedentary Behaviour | Past seven days
  Average weekday and weekend domain-specific time spent sedentary over the past 7 days will be assessed through the modified SIT-Q 7d questionnaire. Participants indicate on a scale of responses the range of times that best correspond to the average amount of time they spent sedentary on weekdays/weekends in domains of: Sleeping and Napping, Meals, Transportation, Occupation(s), Screen Time, and Other Activities, during the past 7 days. Response ranges typically span 30 minutes to 1 hour (e.g., Less than 30 minutes, 1-2 hours).
  Average total sitting time per weekday will be assessed through a single question on the International Physical Activity Questionnaire Seven - Short Form Past 7 Days (IPAQ-S7S): "During the last 7 days, how much time did you spend sitting on a weekday?"
Depression | Past seven days
  Depressive symptomatology will be assessed through the Centre for Epidemiological Studies Depression Scale (CES-D).
  The CES-D scale is a short self-report scale designed to measure depressive symptomatology in the general population. Participants indicate how often in the past week they have felt or behaved for each of the 20 feelings/behaviors in the scale. Options range from: rarely or none of the time (less than 1 day), some or little of the time (1-2 days), occasionally or a moderate amount of time (3-5 days), and most or all of the time (5-7 days). These options correspond to a score of either: 0, 1, 2, or 3, depending on the framing of the question.
  A total score is achieved through summing the scores for all 20 questions; scores range from 0-60, with lower scores indicating a lower symptomatomology for depression. A clinical cut-off point of 20 has been recommended.
Anxiety (State) | Baseline
  State anxiety will be assessed through the State-Trait Anxiety Inventory (STAI) Form Y-1. Participants read each of the 20 statements and then write the number in the blank at the end of the statement that indicates how they feel right now (i.e., at this moment).
  Responses range from: 1 - not at all, to 4 - very much so; these response correspond to a score of 1-4 for anxiety-related items, and 4-1 for anxiety-absent items. A total score is obtained by summing the scores for each question. Total scores range from 20-80, with higher scores indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the State Anxiety scale.

OTHER OUTCOMES:
Age | Baseline
  Assessed with a single-item question: "What is your age?"
Gender | Baseline
  Assessed with a single-item question: "What is your preferred gender?"
Program of study | Baseline
  Assessed with a single-item question: "What is your current program of study?"
Year of study | Baseline
  Assessed with a single-item question: "What is your current year of study?"
Degree Pursuing | Baseline
  Assessed with a single-item question: "What degree are you pursuing?"
Ethnicity | Baseline
  Assessed with a single-item question: "Which ethnicity do you most closely identify with?"

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, PhD, Principal Investigator — Western University
Locations (1):
- Exercise and Health Psychology Lab, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of the research results, IPD will be shared into the Federated Research Data Repository (FRDR)
Supporting Information: Study Protocol
Time Frame: Data will become available upon publication of the research results, and will be available for 5 years after depositing.
Access Criteria: Members of the FRDR will be able to access the data.
URL: http://www.frdr.ca/repo/?locale=en

REFERENCES:
- [Background] Wijndaele K, DE Bourdeaudhuij I, Godino JG, Lynch BM, Griffin SJ, Westgate K, Brage S. Reliability and validity of a domain-specific last 7-d sedentary time questionnaire. Med Sci Sports Exerc. 2014 Jun;46(6):1248-60. doi: 10.1249/MSS.0000000000000214. PMID 24492633
- [Background] Sui W, Prapavessis H. Standing Up for Student Health: An Application of the Health Action Process Approach for Reducing Student Sedentary Behavior-Randomised Control Pilot Trial. Appl Psychol Health Well Being. 2018 Mar;10(1):87-107. doi: 10.1111/aphw.12105. Epub 2017 Dec 5. PMID 29205909
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Ryan RM, Frederick C. On energy, personality, and health: subjective vitality as a dynamic reflection of well-being. J Pers. 1997 Sep;65(3):529-65. doi: 10.1111/j.1467-6494.1997.tb00326.x. PMID 9327588
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Vilagut G, Forero CG, Barbaglia G, Alonso J. Screening for Depression in the General Population with the Center for Epidemiologic Studies Depression (CES-D): A Systematic Review with Meta-Analysis. PLoS One. 2016 May 16;11(5):e0155431. doi: 10.1371/journal.pone.0155431. eCollection 2016. PMID 27182821
- [Background] Radloff LS: The CES-D Scale: a self-report depression scale for research in the general population. Applied Psychological Measurement 1:385-401, 1977.
- See also: SoSci Survey website - host of electronic questionnaire — http://soscisurvey.de